CLINICAL TRIAL: NCT03734575
Title: Prospective, Multi-Center Study of the ClariCore Optical Biopsy System in Patients Undergoing Transperineal Prostate Biopsy for Prostate Tissue Classification Algorithm Development
Brief Title: ClariCore System Used in Transperineal Prostate Biopsy
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Company funding
Sponsor: Precision Biopsy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CIP-1012
Record Dates: First submitted 2018-10-16; First posted 2018-11-08 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- ClariCore System (Experimental): Biopsy tissue, correlative spectral data, T2-weighted MR scans and ultrasound images acquired with the ClariCore System will be collected and recorded during standard practice transperineal biopsy.
  Interventions: Device: ClariCore System

INTERVENTIONS:
Device: ClariCore System — The user will perform a standard trans-perineal biopsy and collect a number of biopsy cores as per standard practice.

SUMMARY:
The overall objective of this study is to acquire ultrasound images, spectral data and prostate tissue biopsy cores using the ClariCore System via a transperineal approach.

DETAILED DESCRIPTION:
The overall objective of this study is to acquire ultrasound images, spectral data and prostate tissue biopsy cores using the ClariCore System via a transperineal approach. Ultrasound images corresponding to each needle insertion and T2-weighted MR scans will be saved for the purpose of further algorithm development that will provide physicians with real time tissue classification in conjunction with location information from the ultrasound imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Males per Investigator assessment appropriate for transperineal prostate biopsy
2. Patient scheduled for transperineal prostate biopsy based on standard of care urologic requirements to assess for tissue malignancy
3. Prostate volume > 20cc and length at least 22mm as verified by ultrasound or prostate MRI prior to the procedure
4. Patient must be able to provide legal consent and signs an IRB (Institutional Review Board)/EC (Ethics Committee) approved Informed Consent form to participate in the study prior to any study mandated determinations or procedure

Exclusion Criteria:

1. Any anatomical or co-morbidity contraindications to transperineal prostate biopsy or transperineal prostate mapping biopsy
2. Acute painful perianal disorder (i.e. rectal abscess)
3. Symptomatic, acute prostatitis
4. Surgical absence of a rectum or the presence of a rectal fistula
5. Patient has systemic infection or evidence of any surgical site infection (superficial or organ space), including active urinary tract infection
6. Previous prostate intervention [TURP (bipolar, monopolar, laser)] TUMT, HIFU, Cryo, Rezum, Urolift], not including previous prostate biopsy
7. Current required use of blood thinning agents for medical comorbidity which prohibits the cessation of use as typically required per standard of care (SOC) prior to a medical procedure; or history of a bleeding disorder (e.g. coagulopathy)
8. Prior pelvic irradiation
9. Actively receiving therapy for the treatment of cancer (except for patients on 5-alpha reductase inhibitors, or non-melanoma skin cancers that are managed nonsystemically)
10. Actively receiving intravesical therapy or within 6 months of treatment for bladder cancer
11. Patient has compromised immune system, in the opinion of the Investigator
12. Active inflammatory bowel disease within the last 6 months
13. Any condition, or history of illness or surgery that, in the opinion of the Investigator, might confound the results of the study or pose additional risks to the patient (e.g.

    significant cardiovascular conditions or allergies)
14. Patient is not likely to comply with the protocol or follow up evaluation
15. Patient is participating in a clinical trial of another investigational drug or device that may impact participation in this clinical study

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Males per Investigator assessment appropriate for transperineal prostate biopsy
Enrollment: 60 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-09 (Estimated)

PRIMARY OUTCOMES:
Correlation of histopathology of tissue with ultrasound images and spectral data | At time of procedure
  The correlation of histopathology of tissue biopsy core samples with the corresponding spectral data and ultrasound images obtained in vivo for the purpose of tissue classification algorithm development using a transperineal approach.

SECONDARY OUTCOMES:
Incidence of Adverse Events (Safety) | At time of procedure
  The cumulative incidence of adverse events related to the device or the procedure. The cumulative incidence of serious adverse events (SAEs) related to the device or the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: James Wysock, MD, Principal Investigator — NYU Langone Urology Associates
Locations (2):
- United States (2):
  - The James Buchanan Brady Urological Institute and Department of Urology, Baltimore, Maryland
  - NYU Langone Urology Associates, New York, New York

IPD SHARING:
Plan to Share IPD: No